CLINICAL TRIAL: NCT00441961
Title: Treatment With High Dose Methotrexate in Patients With Eosinophilic Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: H. Knaapen, MD, Radboud University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mtx in eosinophilic fasciitis
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2010-07

CONDITIONS: Fasciitis
Keywords: Eosinophilic fasciitis, Shulman's syndrome, methotrexate
MeSH Terms: conditions — Fasciitis; Eosinophilic Fasciitis | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: methotrexate — methotrexate

SUMMARY:
Evaluate the effect of high dose MTX on skin induration in patients with eosinophilic fascia.

DETAILED DESCRIPTION:
Eosinophilic fasciitis (EF)is a fibrosing skin disorder extensively involving the deep fascia. The aim of this pilot study is to evaluate the effect of high dose MTX on skin induration in patients with EF. In addition, we study the effect of this treatment on joint mobility, peripheral blood eosinophilia, functional ability, and pulmonary function. By administering high dose MTX intravenously every four weeks with a Leukovorin rescue, we hope to induce a more pronounced and sustained effect on the involved skin with less (long-lasting) side effects.

ELIGIBILITY:
Inclusion Criteria:

* Eosinophilic fasciitis as defined by clinical judgement of an expert,
* Histologically confirmed with a skin-fascia-muscle biopsy, and in additon:

  * Either the presence of a modified skin score according to Zachariae of 8 or higher (0-18), regarded as a generalised eosinophilic fasciitis or the presence of severe contractures due to eosinophilic fasciitis lesions.

Exclusion Criteria:

* Age < 18 yrs
* Contraindications to MTX: AST/ALT level > 2 times upper limit of normal, WBC count < 3.5 x 109/l or platelet count < 150 x 109/l, serum creatinine > 130 micromol/l or clearance < 50 ml/min, confirmed by two repeated tests within one month.
* Chronic liver disease, insulin dependant diabetes mellitus, alcohol abuse
* Restrictive pulmonary disease (total lung capacity or vital capacity < 40% of predicted) or interstitial lung disease (KCO < 60% of predicted)
* Pregnancy or child bearing potential without adequate contraception
* The presence of any serious co-morbidity or malignancy
* Use of other anti-folate drugs than MTX

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-10; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Efficacy is evaluated after 6 months. | December 2008

CONTACTS AND LOCATIONS:
Overall Officials: H. Knaapen, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] Mertens JS, Zweers MC, Kievit W, Knaapen HK, Gerritsen M, Radstake TR, van den Hoogen FH, Creemers MC, de Jong EM. High-Dose Intravenous Pulse Methotrexate in Patients With Eosinophilic Fasciitis. JAMA Dermatol. 2016 Nov 1;152(11):1262-1265. doi: 10.1001/jamadermatol.2016.2873. PMID 27541801